CLINICAL TRIAL: NCT01844895
Title: Substudy-A Phase IIIB Multicenter, Randomized, Double-Blind, Double-Dummy Study to Compare the Efficacy and Safety of Abatacept Administered Subcutaneously and Intravenously in Subjects With Rheumatoid Arthritis, Receiving Background Methotrexate, and Experiencing an Inadequate Response to Methotrexate
Brief Title: Methotrexate-Inadequate Response Autoinjector Device Sub Study
Acronym: MTX-IR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM101-174 Substudy-2; 2007-005434-37 (EudraCT Number)
Record Dates: First submitted 2013-04-05; First posted 2013-05-03 (Estimated); Results first posted 2015-07-01 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abatacept (Autoinjector and Prefilled Syringe) (Experimental): Abatacept (prefilled syringe) 125 mg/device solution subcutaneously weekly for 3 months
  Abatacept (autoinjector) 125 mg/device solution subcutaneously weekly for 1 month
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept
  Other Names: Orencia; BMS-188667

SUMMARY:
The purpose of this study is to implement a substudy in approximately 120 rheumatoid arthritis (RA) subjects to compare the steady-state serum trough concentration (Cminss), Cmax and area under the curve (AUC) during the dosing interval (TAU) of subcutaneous (SC) Abatacept injection of 125 mg via the autoinjector and via the BD Hypak™ Physiolis prefilled syringe.

DETAILED DESCRIPTION:
Study Classification:

* Safety: show if the drug is safe under conditions of proposed use
* Efficacy: measure of an intervention's influence on a disease or health condition
* Safety/Efficacy
* Pharmacokinetics: the action of a drug in the body over a period of time including the process of absorption, distribution and localization in tissue, biotransformation, and excretion of the compound.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects who have been treated in the long term (LT) with open-label SC Abatacept for at least 3 months
* Must continue to meet inclusion criteria specified in main IM101-174 Study Protocol

Exclusion Criteria:

* Participation in previous device substudy (implemented by Amendment 10)
* Must continue to meet exclusion criteria specified in main IM101-174 Study Protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Autoinjector Substudy initiated April 2013; completed July 2014. Those participating in the long term main (parent) study IM101-174 who received weekly open-label SC 125mg abatacept injections via prefilled syringe for at least 3 months and who did not participate in a previous device substudy were eligible to enroll in the autoinjector substudy.
Groups:
- 125 mg Abatacept (Autoinjector and Prefilled Syringe): 125 mg SC abatacept was self administered weekly via pre-filled syringes from Day 1 up to Day 29 when the participant was switched to self administering 125 mg SC abatacept via the autoinjector device for 3 months. Participants could discontinue from the autoinjector substudy and switch back to prefilled syringes at any time during the study. Following the 4 months of the substudy, participants could continue to receive abatacept SC via the autoinjector or switch back to the prefilled syringe until the close of the IM101-174 parent study.
Period: Day 1 to Day 28 - Pre-filled Syringe
Arm/Group | 125 mg Abatacept (Autoinjector and Prefilled Syringe)
Started | 120
Completed | 117
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Clinic Closed | 1
Period: Day 29 - Day113 - Autoinjector
Arm/Group | 125 mg Abatacept (Autoinjector and Prefilled Syringe)
Started | 117
Completed | 111
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Difficulty using device | 3
Not completed — planned surgery | 1

BASELINE CHARACTERISTICS:
Population: The Treated Analysis population included all enrolled participants who received at least 1 dose of study medication administered with the autoinjector during the substudy period.
Groups:
- 125 mg Abatacept (Autoinjector and Prefilled Syringe): Participants self administered 125 mg SC abatacept weekly via prefilled syringe from Day 1 up to Day 29. Starting on Day 29, 125 mg SC abatacept was self administered weekly via autoinjector for 3 months.
Arm/Group | 125 mg Abatacept (Autoinjector and Prefilled Syringe)
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 17
Region of Enrollment [Number; unit: participants]
  South America | 100
  North America | 17
Body Weight [Number; unit: participants]
  <60 kilogram (kg) | 28
  60 - 100 kg | 83
  >100 kg | 6
Duration of Disease [Median (Full Range); unit: years] | 6.0 [0 to 41.0]
Methotrexate (MTX) Dose at SubStudy Baseline [Mean (Standard Deviation); unit: mg/wk] — Substudy baseline=Day 1 of Substudy. MTX dose is measured in milligrams per week (mg/wk).
  mg/wk | 17.0 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Analysis: Adjusted Geometric Mean Observed Serum Trough Concentration at Steady State (Cminss) of Abatacept Using a Prefilled Syringe (Measured on Day 29) and Using an Autoinjector (Measured on Day 113)
Description: Abatacept SC was self-administered with a prefilled syringe every 7 days for the first 4 weeks until Day 29; Blood samples for PK were taken pre-dose (0 hour) on Days 29 and 113. Serum concentrations of abatacept were analyzed using a validated enzyme-linked immunosorbent assay (ELISA). Steady-state trough observed concentration in serum (Cminss) was measured in micrograms/milliliter (μg/mL). Adjusted geometric mean and 90% confidence interval (CI) are presented.
Time Frame: Day 29, Day 113
Population: The primary PK analysis population is a subset of the Treated Analysis population with (1) viable Cmin data on both substudy Days 29 and 113 (2) no missed Abatacept dose during the substudy period.
Measure: Geometric Mean (90% Confidence Interval); unit: μg/mL
Groups:
- 125 mg Abatacept SC Using Prefilled Syringe - Day 29: 125 mg Abatacept SC was self-administered with a BD Hypak™ Physiolis prefilled syringe every 7 days for the first 4 weeks of the substudy until Day 29.
- 125 mg Abatacept SC Using Autoinjector - Day 113: 125 mg Abatacept SC was self-administered with an autoinjector starting on Day 29. Participants continued to self-administer abatacept with the autoinjector every 7 days for 3 months.
Arm/Group | 125 mg Abatacept SC Using Prefilled Syringe - Day 29 | 125 mg Abatacept SC Using Autoinjector - Day 113
Number analyzed (Participants) | 88 | 88
μg/mL | 27.76 [24.44 to 31.53] | 25.32 [22.59 to 28.38]
Statistical Analysis 1: Comparison: 125 mg Abatacept SC Using Prefilled Syringe - Day 29 vs 125 mg Abatacept SC Using Autoinjector - Day 113; A mixed-effect model of log (Cminss) with device and substudy baseline weight category (< 60 kg,60-100 kg, > 100 kg) as fixed effects and participant as a random effect was used. Point estimates and 90% CIs for device differences on the log scale were exponentiated to obtain estimates for ratios of geometric means on the original scale. No adjustment was made for multiplicity. PK comparability was concluded if the 90% CIs for the ratios of geometric means were contained within 80% to 125%; Test type: Superiority or Other; geometric mean ratio = 0.91, 90% CI 2-sided [0.83 to 1.00]

2. Secondary Outcome: PK Analysis: Geometric Mean of Maximum Observed Serum Concentration (Cmax) of Abatacept During the Sampling Period Between Substudy Days 22 and 29 for the Prefilled Syringe and Between Substudy Days 106 and Day 113 for the Autoinjector
Description: Abatacept SC was self-administered with a BD Hypak™ Physiolis prefilled syringe every 7 days for the first 4 weeks of the substudy until Day 29; Blood samples for PK were taken on Days 1 and 22 at 0 hour (predose), Day 24 at 48 hour (h) post dose, Day 25 at 72 h post dose, Day 26 at 96 h post dose and Day 29 at 0 h (predose). On substudy Day 29, participants were switched from the prefilled syringe to the autoinjector. Participants continued to self-administer abatacept with the autoinjector every 7 days following Day 29 for the remaining 3 months of the substudy; Blood samples for PK were taken on Day 108 at 48 h post dose, Day 109 at 72 h post dose, Day 110 at 96 h post dose and at Day 113 0h (predose). Serum concentrations of abatacept were analyzed using a validated ELISA. Cmax was measured in μg/mL.
Time Frame: Days 22, 24, 25, 26, 29 (prefilled syringe); Days 106, 108, 109, 110, 113 (autoinjector)
Population: PK population: A subset of the treated population with at least 1 PK sample collected/assessed for serum concentration after start of autoinjector. Participants did not miss either 0-hour or 168-hour samples and not missed 2 or more time points in the PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- 125 mg Abatacept SC Prefilled Syringe - Days 22, 24, 25, 26,29: 125 mg Abatacept SC was self-administered with a BD Hypak™ Physiolis prefilled syringe every 7 days for the first 4 weeks of the substudy until Day 29.
- 125 mg Abatacept SC Autoinjector-Days 106, 108, 109, 110, 113: 125 mg Abatacept SC was self-administered with a autoinjector starting on Day 29. Participants continued to self-administer abatacept with the autoinjector every 7 days for 3 months.
Arm/Group | 125 mg Abatacept SC Prefilled Syringe - Days 22, 24, 25, 26,29 | 125 mg Abatacept SC Autoinjector-Days 106, 108, 109, 110, 113
Number analyzed (Participants) | 95 | 78
μg/mL | 40.9 (48) | 39.8 (58)

3. Secondary Outcome: PK Analysis: Median Time to Achieve Cmax (Tmax) During the Sampling Period Between Days 22 and 29 for the Prefilled Syringe and Between Days 106 and Day 113 for the Autoinjector
Description: Abatacept SC was self-administered with a BD Hypak™ Physiolis prefilled syringe every 7 days for the first 4 weeks of the substudy until Day 29; Blood samples for PK were taken on Days 1 and 22 at 0 hour (predose), Day 24 at 48 hour (h) post dose, Day 25 at 72 h post dose, Day 26 at 96 h post dose and Day 29 at 0 h (predose). On substudy Day 29, participants were switched from the prefilled syringe to the autoinjector. Participants continued to self-administer abatacept with the autoinjector every 7 days following Day 29 for the remaining 3 months of the substudy; Blood samples for PK were taken on Day 108 at 48 h post dose, Day 109 at 72 h post dose, Day 110 at 96 h post dose and at Day 113 0h (predose). Serum concentrations of abatacept were analyzed using a validated ELISA. Tmax was measured in hours (h).
Time Frame: Days 22, 24, 25, 26, 29 (prefilled syringe); Days 106, 108, 109, 110,113 (autoinjector)
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Groups:
- 125 mg Abatacept SC Prefilled Syringe-Days 22, 24, 25, 26, 29: 125 mg Abatacept SC was self-administered with a BD Hypak™ Physiolis prefilled syringe every 7 days for the first 4 weeks of the substudy until Day 29.
Arm/Group | 125 mg Abatacept SC Prefilled Syringe-Days 22, 24, 25, 26, 29 | 125 mg Abatacept SC Autoinjector-Days 106, 108, 109, 110, 113
Number analyzed (Participants) | 95 | 78
h | 70.00 [0 to 168.7] | 56.34 [0 to 171.1]

4. Secondary Outcome: Geometric Mean of Area Under Serum Concentration-time (AUC) During a Dosing Interval (TAU) of Abatacept During the Sampling Period Between Days 22 and 29 for the Prefilled Syringe and Between Days 106 and Day 113 for the Autoinjector
Description: Abatacept SC was self-administered with a BD Hypak™ Physiolis prefilled syringe every 7 days for the first 4 weeks of the substudy until Day 29; Blood samples for PK were taken on Days 1 and 22 at 0 hour (predose), Day 24 at 48 hour (h) post dose, Day 25 at 72 h post dose, Day 26 at 96 h post dose and Day 29 at 0 h (predose). On substudy Day 29, participants were switched from the prefilled syringe to the autoinjector. Participants continued to self-administer abatacept with the autoinjector every 7 days following Day 29 for the remaining 3 months of the substudy; Blood samples for PK were taken on Day 106 at 0 h (predose), Day 108 at 48 h post dose, Day 109 at 72 h post dose, Day 110 at 96 h post dose and at Day 113 0h (predose). Serum concentrations of abatacept were analyzed using a validated ELISA. AUC(TAU) where TAU = 168 hours was calculated in µg*h/mL
Time Frame: Days 22, 24, 25, 26,29 (prefilled syringe); Days 106, 108, 109, 110, 113 (autoinjector)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | 125 mg Abatacept SC Prefilled Syringe-Days 22, 24, 25, 26, 29 | 125 mg Abatacept SC Autoinjector-Days 106, 108, 109, 110, 113
Number analyzed (Participants) | 95 | 78
µg*h/mL | 5740 (47) | 5643 (50)

5. Secondary Outcome: Geometric Mean of Trough Serum Concentration (Cmin) Over Time and During the Switch From Prefilled Syringe to Autoinjector on Days 22, 29, 57, 85, 106, and 113
Description: Abatacept SC was self-administered with a BD Hypak™ Physiolis prefilled syringe every 7 days for the first 4 weeks of the substudy until Day 29; Blood samples for PK were taken at 0 hour (predose). On substudy Day 29, participants were switched from the prefilled syringe to the autoinjector. Participants continued to self-administer abatacept with the autoinjector every 7 days following Day 29 for the remaining 3 months of the substudy. Blood samples for PK were taken at 0 hour (predose). Serum concentrations of abatacept were analyzed using a validated ELISA. Steady-state trough observed concentration in serum (Cminss) was measured in micrograms/milliliter (μg/mL).
Time Frame: Days 22, 29, 57, 85, 106, and 113
Population: PK population: A subset of the treated population with at least 1 PK sample collected/assessed for serum concentration after start of autoinjector and with Cmin obtained appropriately (7 days + or -3 days after the previous dose).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- 125 mg Abatacept SC Using Prefilled Syringe: 125 mg Abatacept SC was self-administered with a BD Hypak™ Physiolis prefilled syringe every 7 days for the first 4 weeks of the substudy until Day 29.
- 125 mg Abatacept SC Using Autoinjector: 125 mg Abatacept SC was self-administered with a autoinjector starting on Day 29. Participants continued to self-administer abatacept with the autoinjector every 7 days throughout the substudy.
Arm/Group | 125 mg Abatacept SC Using Prefilled Syringe | 125 mg Abatacept SC Using Autoinjector
Number analyzed (Participants) | 108 | 105
μg/mL
  Day 22 (n=104, 0) Pre-filled Syringe Only | 29.09 (48) | NA (NA) — n=0 for autoinjector on Days 22 and 29
  Day 29 (n=108, 0) Pre-filled Syringe Only | 30.58 (51) | NA (NA) — n=0 for autoinjector on Days 22 and 29
  Day 57 (n=0,105) Autoinjector Only | NA (NA) — n=0 for prefilled syringe after Day 29 | 28.79 (59)
  Day 85 (n=0,104) Autoinjector Only | NA (NA) — n=0 for prefilled syringe after Day 29 | 25.73 (53)
  Day 106 (n=0, 91) Autoinjector Only | NA (NA) — n=0 for prefilled syringe after Day 29 | 30.42 (56)
  Day 113 (n=0,100) Autoinjector Only | NA (NA) — n=0 for prefilled syringe after Day 29 | 28.06 (51)

6. Secondary Outcome: Number of Participants With Positive Anti-Abatacept or Anti-CTLA4 Antibody Responses by Electrochemiluminescence (ECL) on Day 29 and Day 113.
Description: Serum samples for immunogenicity were evaluated for presence of anti-abatacept antibodies using a validated bridging ECL on Day 29 and Day 113. The ECL assay differentiated between 2 antibody specificities: the immunoglobulin (Ig) G and/or junction region and cytotoxic leukocyte antigen 4 (CTLA4) and possibly Ig. A positive immunogenicity response relative to baseline was defined as: A missing baseline immunogenicity measurement and a positive analytical laboratory reported immunogenicity response post-baseline; A negative baseline immunogenicity response and a positive analytical laboratory reported immunogenicity response post-baseline; A positive baseline immunogenicity response and a positive analytical laboratory reported immunogenicity response post-baseline that has a titer value strictly greater than the baseline titer value.
Time Frame: Days 29 and 113
Population: A subset of the treated analysis population for whom at least 1 immunogenicity sample was collected and assessed for serum anti-abatacept antibodies, were summarized.
Measure: Number; unit: participants
Groups:
- 125 mg Abatacept SC Prefilled Syringe - Day 29: 125 mg Abatacept SC was self-administered with a BD Hypak™ Physiolis prefilled syringe every 7 days for the first 4 weeks of the substudy until Day 29.
- 125 mg Abatacept SC Autoinjector- Day 113: 125 mg Abatacept SC was self-administered with a autoinjector starting on Day 29. Participants continued to self-administer abatacept with the autoinjector every 7 days throughout the substudy.
Arm/Group | 125 mg Abatacept SC Prefilled Syringe - Day 29 | 125 mg Abatacept SC Autoinjector- Day 113
Number analyzed (Participants) | 115 | 103
participants
  CTLA4 and Possibly Ig | 1 | 1
  Ig and/or Junction | 5 | 2

ADVERSE EVENTS:
Time Frame: Day 1 of the substudy up to 56 days post the last autoinjector dose.
Description: Substudy was approximately 4 months in length. Participants on Day 1 up to Day 29 used prefilled syringes to self administer study drug and then starting Day 29 and for 3 additional months, participants used an autoinjector to self administer study drug.
Groups:
- Abatacept Via Autoinjector Only (Day 29 to End of Study): Participants received 125 mg SC abatacept via the autoinjector starting Day 29 and through the remaining 3 months of the substudy.
- Abatacept Cumulative (Prefilled Syringe and Autoinjector): 125 mg SC abatacept was self administered weekly via pre-filled syringes from Day 1 up to Day 29 when the participant was switched to self administering 125 mg SC abatacept via the autoinjector device for 3 months.
Arm/Group | Abatacept Via Autoinjector Only (Day 29 to End of Study) | Abatacept Cumulative (Prefilled Syringe and Autoinjector)
Serious Adverse Events (participants affected / at risk) | 3/117 | 3/117
Other Adverse Events (participants affected / at risk) | 40/117 | 43/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept Via Autoinjector Only (Day 29 to End of Study) (N=117) | Abatacept Cumulative (Prefilled Syringe and Autoinjector) (N=117)
HiNI Influenza (Infections and infestations) | 1 | 1
Postoperative wound infection (Infections and infestations) | 1 | 1
Myocardial Ischemia (Cardiac disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept Via Autoinjector Only (Day 29 to End of Study) (N=117) | Abatacept Cumulative (Prefilled Syringe and Autoinjector) (N=117)
Nasopharyngitis (Infections and infestations) | 7 | 9
Pharyngitis (Infections and infestations) | 5 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 6
Bronchitis (Infections and infestations) | 2 | 3
Hypertension (Vascular disorders) | 2 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Conjunctivitis (Infections and infestations) | 1 | 1
Ear Infection (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 1 | 1
Impetigo (Infections and infestations) | 1 | 1
Pharyngitis Bacterial (Infections and infestations) | 1 | 1
Post Procedural Infection (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 1 | 1
Vaginal Infection (Infections and infestations) | 1 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Plantar Fascitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Irritable Bowel syndrome (Gastrointestinal disorders) | 0 | 1
Drug intolerance (General disorders) | 0 | 1
Injection site Hemorrhage (General disorders) | 1 | 1
Injection site pruritus (General disorders) | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 1
Blood Pressure Increased (Investigations) | 0 | 1
Transaminases Increased (Investigations) | 1 | 1
Cervical Radiculopathy (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 1
Seasonal Allergy (Immune system disorders) | 1 | 1
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Postmenopausal hemorrhage (Reproductive system and breast disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.